CLINICAL TRIAL: NCT02987101
Title: Treatment of Chronic Leg Ulcers With Autologous Stromal Vascular Fraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Navid Toyserkani, Resident, PhD fellow, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-201502002
Record Dates: First submitted 2016-11-24; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Leg Ulcer
MeSH Terms: conditions — Leg Ulcer | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous SVF + Standard of care (Experimental): local injection around and under wound with autologous stromal vascular fraction.
  Standard wound care is given independent of this study.
  Interventions: Procedure: Liposuction; Other: Standard wound care; Drug: Adipose-Derived Regenerative Cells
- Standard of care (Other): Standard wound care is given independent of this study.
  Interventions: Other: Standard wound care

INTERVENTIONS:
Procedure: Liposuction — Adipose tissue is harvested by liposuction from either abdomen or thighs.
  Arms: Autologous SVF + Standard of care
Other: Standard wound care — Patients will receive standard wound care and dressings independent of their participation in this study at the discretion of the wound nurses.
Drug: Adipose-Derived Regenerative Cells — Cells isolated from adipose-derived tissue will be injected locally around and under the wound.
  Arms: Autologous SVF + Standard of care

SUMMARY:
Chronic leg ulcers are associated with decreased quality of life and an increased mortality. In many cases these ulcers are treated conservatively and the healing time can be several months. In this open randomized clinical trial we will examine if we can accelerate wound healing when using autologous stromal vascular fraction as an adjunct to standard wound care.

DETAILED DESCRIPTION:
Chronic leg ulcers are associated with decreased quality of life and an increased mortality. In many cases these ulcers are treated conservatively and the healing time can be several months. In this open randomized clinical trial we will examine if we can accelerate wound healing when using autologous stromal vascular fraction (SVF) as an adjunct to standard wound care.

The plan is to include 30 patients with arterial or arteriovenous chronic leg ulcers and these are randomized in two groups of which one receives standard wound care only and the other group receives autologous stromal vascular fraction treatment in addition to standard wound care.

ELIGIBILITY:
Inclusion Criteria:

* Arteriovenous chronic leg ulcer
* Present beyond 4 months
* Conservative treatment not leading to progress
* Wound size between 2-30cm2
* ankle-brachial index (ABI) ( 50-90% and/or toe pressure 50-70% and where ankle pressure > 60 mmHg or toe pressure > 40 mmHg
* Written informed consent

Exclusion Criteria:

* Uncontrolled wound infection
* Osteomyelitis
* Hemoglobin <6.0mmol/L
* HbA1c >80mmol/mol
* Underlying malignancy
* Pregnancy or lactating
* Renal insufficiency requiring dialysis
* Charcot foot
* Underlying malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in wound size | 6 months
  Photography is taken every 2 weeks until complete wound healing. Final follow-up date regardless of complete wound healing or not is 6 months.

SECONDARY OUTCOMES:
Distal blood pressure measurement | 6 months
  Change in distal blood pressure measurement before and 6 months after treatment
Transcutaneous oxygen tension | 6 months
  Change in transcutaneous oxygen tension around the wound before and 6 months after treatment.
Treatment-related adverse events | 6 months
  Monitoring of any side effects or complications related to intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jens A Sørensen, MD PhD, Study Chair — Dept. Plastic Surgery, OUH, Consultant, Professor
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided